CLINICAL TRIAL: NCT01635881
Title: EMERGE: Evaluation of Coronary Luminal Diameter Enlargement With Emerge™ 1.20 mm Percutaneous Transluminal Coronary Angioplasty (PTCA) Dilatation Catheter
Brief Title: Evaluation of Coronary Luminal Diameter Enlargement With Emerge™ 1.20 mm PTCA Dilatation Catheter
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S2228
Record Dates: First submitted 2012-05-25; First posted 2012-07-10 (Estimated); Results first posted 2013-11-06 (Estimated); Last update posted 2013-11-06 (Estimated); Status verified 2013-10

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Emerge (Experimental): Single arm with investigational Emerge™ 1.20 mm PTCA Dilatation Catheter
  Interventions: Device: Emerge™ 1.20 mm PTCA Dilatation Catheter

INTERVENTIONS:
Device: Emerge™ 1.20 mm PTCA Dilatation Catheter — The Emerge 1.20 mm device is the next-generation Boston Scientific PTCA dilatation catheter. It is a sterile, single-use, intravascular medical device used to improve lumen diameter.
  The catheter consists of a shaft with a balloon near the distal tip. The balloon is designed to provide an inflatable segment of known diameter and length at recommended pressures.

SUMMARY:
To evaluate the acute safety and device procedural success of the Emerge 1.20 mm PTCA dilatation catheter when used as a pre-dilatation device in the stenotic portion of coronary arteries or bypass grafts.

ELIGIBILITY:
Clinical Inclusion Criteria:

1. Subject is ≥ 18 years of age.
2. Subject or a legally authorized representative must provide written informed consent prior to any study related procedures.
3. Subject must agree not to participate in any other clinical study during hospitalization for the index procedure.
4. Subjects must have a single or double vessel coronary artery disease and clinical evidence of ischemic heart disease, such as stable / unstable angina or silent ischemia.

Angiographic Inclusion Criteria:

1. Subject must have de novo or restenotic lesion(s) in native coronary arteries or bypass grafts that are suitable for percutaneous coronary intervention. An embolic protection device must be used in all Saphenous venous grafts (SVG) interventions performed during the index procedure.
2. A maximum of two lesions, including at least one target lesion, in up to two coronary arteries.
3. Target and non-target lesions must be located in different coronary arteries or bypass grafts.
4. Target lesion(s) must have a diameter stenosis of ≥70% by visual estimation and may include chronic total occlusions (CTO)
5. Treatment of non-target lesion, if any, must be completed prior to treatment of target lesion and must be deemed a clinical angiographic success.

Exclusion Criteria:

1. Subject with a known hypersensitivity or contraindication to Aspirin, Heparin, Bivalirudin, anti-platelet medications, or sensitivity to contrast media which cannot be adequately pre-medicated.
2. Subject with known diagnosis of an acute myocardial infarction (AMI) within 72 hours prior to index procedure.
3. Subject with known pregnancy or is nursing. Women of childbearing potential should have a documented negative pregnancy test within 7 days before index procedure.
4. Planned or actual target lesion treatment with an unapproved device, atherectomy, laser, cutting balloon or thrombectomy during the index procedure.
5. A serum creatinine level > 2.0 mg/dl within seven days prior to index procedure.
6. Cerebrovascular accident (CVA) within the past 6 months.
7. Active peptic ulcer or active gastrointestinal (GI) bleeding within the past 6 months.
8. Subject has a known left ventricular ejection fraction (LVEF) <30% (LVEF may be obtained at the time of the index procedure if the value is unknown, if necessary).

Angiographic Exclusion Criteria

1. More than two lesions requiring treatment.
2. Unprotected left main coronary artery disease.
3. Coronary artery spasm of the target vessel in the absence of a significant stenosis.
4. Target lesion with angiographic presence of probable or definite thrombus.
5. Untreated lesions with >50% diameter stenosis remaining in any coronary artery.
6. Target lesion involves a bifurcation requiring treatment with more than one stent or pre-dilatation of a side branch >2.0 mm in diameter.
7. Non-target lesion to be treated during the index procedure meets any of the following criteria:

   1. Located within a bypass graft (venous or arterial)
   2. Left main location
   3. Chronic total occlusion
   4. Involves a bifurcation (e.g., bifurcations requiring treatment with more than 1 stent)
   5. Treatment not deemed a clinical angiographic success

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-07; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David E Kandzari, MD, Principal Investigator — Director, Interventional Cardiology, Chief Scientific Officer, Piedmont Heart Institute
Locations (1):
- Piedmont Heart Institute, Atlanta, Georgia, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment of subjects for EMERGE study started on July 09, 2012 and completed on December 14, 2012. Subjects were recruited at 3 investigational centers.
Groups:
- Emerge: Single arm with investigational Emerge™ 1.20 mm percutaneous transluminal coronary angioplasty (PTCA) Dilatation Catheter
Period: Overall Study
Arm/Group | Emerge
Started | 60
Completed | 60
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Emerge
Number analyzed (Participants) | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 41
  >=65 years | 19
Age Continuous [Mean (Standard Deviation); unit: years] | 60.9 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 43
Race/Ethnicity, Customized [Number; unit: Participants]
  American Indian or Alaska native | 0
  Asian | 0
  Black, or African American | 3
  White | 57
  Hispanic | 0
  Native Hawaiian or Other Pacific Islander | 0
Region of Enrollment [Number; unit: participants]
  United States | 60
Cardiac History [Number; unit: Participants] — More than one Cardiac History measure may be reported for each participant.
  Participants
    Previous Percutaneous Coronary Intervention | 37
    Previous Coronary Artery Bypass Graft | 11
    Previous Myocardial Infarction | 14
    Congestive Heart Failure | 2
    Stable Angina | 24
    Unstable Angina | 25
    Silent Ischemia | 7
Cardiac Risk Factors [Number; unit: Participants] — More than one Cardiac Risk Factor may be reported for each participant.
  Participants
    Smoking, Ever | 36
    Medically Treated Diabetes | 21
    Hyperlipidemia Requiring Medication | 51
    Hypertension Requiring Medication | 56
    Family History of Coronary Artery Disease | 37
Lesion Characteristic: Target Lesion Vessel [Number; unit: Lesions] — Analysis is based on the number of intent-to-treat lesions (n=67).
  Lesions
    Left Anterior Descending Artery | 26
    Circumflex Artery | 14
    Right Coronary Artery | 21
    Left Main Coronary Artery | 1
    Graft | 2
Lesion Characteristic: Lesion Location [Number; unit: Lesions] — Analysis is based on the number of intent-to-treat lesions (n=67).
  Lesions
    Ostial | 11
    Proximal | 16
    Mid | 32
    Distal | 8
Lesion Characteristic: Lesion Length [Number; unit: Lesions] — Analysis is based on the number of intent-to-treat lesions (n=67).
  Lesions
    Less than 18 mm | 51
    From 18 and less than 26 mm | 11
    Greater or equal to 26 mm | 5
Lesion Characteristics [Number; unit: Lesions] — Analysis is based on the number of intent-to-treat lesions (n=67).
  Lesions
    Thrombus | 0
    Tortuosity, Any | 9
    Calcification, Any | 30
    Ulcerated | 0
    Aneurysm | 3
    Intimal Flap | 0
    Total Occlusion | 7
    Eccentric Lesion | 40
Lesion Characteristic: Pre-Procedure Thrombolysis in Myocardial Infarction (TIMI) Flow [Number; unit: Lesions] — Analysis is based on the number of intent-to-treat lesions (n=67).
  Lesions
    0 (no perfusion) | 5
    1 (penetration with minimal perfusion) | 2
    2 (partial perfusion) | 1
    3 (complete perfusion) | 59
Lesion Characteristics [Mean (Standard Deviation); unit: Millimeters] — Analysis is based on the number of intent-to-treat lesions (n=67).
  Millimeters
    Reference Vessel Diameter | 2.6 (0.5)
    Minimum Lumen Diameter | 0.7 (0.4)
    Lesion Length | 15.5 (14.7)
Lesion Characteristic: Percent Diameter Stenosis [Mean (Standard Deviation); unit: Percent Diameter Stenosis] — Analysis is based on the number of intent-to-treat lesions (n=67).
  Percent Diameter Stenosis | 73.0 (12.6)

OUTCOME MEASURES:

1. Primary Outcome: Device Procedural Success
Description: Device procedural success consisting of the following:
  1. Successful delivery, inflation, deflation and withdrawal of the study balloon.
  2. No evidence of vessel perforation, flow limiting dissection (grade C or higher) or reduction in TIMI flow from baseline related to the study balloon.
  3. Final TIMI flow grade of 3 at the conclusion of the percutaneous coronary intervention procedure
Time Frame: Peri-procedural
Population: Analysis population consists of intent-to-treat subject population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Emerge
Number analyzed (Participants) | 60
percentage of participants | 98.3 [91.1 to 100.0]

2. Secondary Outcome: In-hospital Major Adverse Cardiac Events (MACE)
Description: In-hospital MACE:
  1. All death (cardiac and non-cardiac)
  2. Myocardial infarction (MI)
  3. Target Vessel Revascularization (TVR)
  4. In-hospital Stent Thrombosis (ST) within the target vessel
  5. Clinically significant arrhythmias (requiring intervention)
Time Frame: Participants will be followed for the duration of hospital stay (an expected average of 24 hours)
Population: Analysis population consists of intent-to-treat subject population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Emerge
Number analyzed (Participants) | 60
percentage of participants | 6.7 [1.8 to 16.2]

ADVERSE EVENTS:
Time Frame: Serious and non-serious adverse events were collected from the point of subject enrollment through study completion at hospital discharge.
Arm/Group | Emerge
Serious Adverse Events (participants affected / at risk) | 2/60
Other Adverse Events (participants affected / at risk) | 6/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Emerge (N=60)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Haematochrezia (Gastrointestinal disorders) | 1 (1)
Melaena (Gastrointestinal disorders) | 2 (2)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1.0% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Emerge (N=60)
Myocardial infarction (Cardiac disorders) | 3 (3)
Blood creatinine abnormal (Investigations) | 1 (1)
Cardiac enzymes increased (Investigations) | 1 (1)
Urine analysis abnormal (Investigations) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution and Investigator shall have the right to publish the results, provided that before publishing, Institution and Investigator shall submit copies of any proposed publication or presentation to Sponsor for review at least sixty (60) days in advance of submission for publication or presentation to a publisher or other third party. Sponsor reserves the right to delete any confidential information or other proprietary information of Sponsor from the proposed publication or presentation.